CLINICAL TRIAL: NCT03004612
Title: Effect of Linagliptin + Metformin vs Metformin Alone on the Role of Pancreatic Islet Function, Insulin Resistance and Markers of Cardiovascular Risk in Patients With Prediabetes: Randomized Clinical Trial
Brief Title: Effect of Linagliptin + Metformin vs Metformin Alone in Patients With Prediabetes
Acronym: PRELLIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Rodolfo Guardado Mendoza, MDPhD, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEI-22-16
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Prediabetic State; Insulin Resistance
Keywords: prediabetes
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Linagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linagliptin + Metformin plus lifestyle (Experimental): Patients are randomized to receive for 24 months Linagliptin 2.5mg + metformin 850mg every 12 hours. The start of the dose in this group will be gradual so that at the month of treatment the patient can be with the full doses. Together with this, patients will receive a lifestyle modification program seeking to reduce 5-7% of body weigh and increase physical activity to 90-150min/week.
  Interventions: Combination Product: Linagliptin + metformin
- Metformin plus lifestyle (Active Comparator): Patients are randomized to receive for 24 months Metformin 850mg every 12 hours. The start of the dose in this group will be gradual so that at the month of treatment the patient can be with the full doses. Together with this, patients will receive a lifestyle modification program seeking to reduce 5-7% of body weigh and increase physical activity to 90-150min/week.
  Interventions: Drug: Metformin

INTERVENTIONS:
Combination Product: Linagliptin + metformin — Linagliptin-Metformin 2.5/850mg twice daily plus a lifestyle modification program based on nutritional assesment, physical activity prescription and general counseling
  Other Names: Tradjenta Duo
  Arms: Linagliptin + Metformin plus lifestyle
Drug: Metformin — Metformin 850mg twice daily plus a lifestyle modification program based on nutritional assesment, physical activity prescription and general counseling
  Arms: Metformin plus lifestyle

SUMMARY:
Type 2 diabetes is a worldwide epidemic disease, and preventive strategies are needed to face this health problem. The goal of this clinical trial is to evaluate the effect of linagliptin + metformin vs metformin alone on physiopathological parameters, such as glucose metabolism, insulin resistance, insulin secretion and pancreatic beta cell function in patients with impaired fasting glucose plus impaired glucose tolerance, during 24 months.

DETAILED DESCRIPTION:
The main goal of this clinical trial is to compare the effect of two different treatments during 24 months:

1. Lifestyle modification program + metformin 850mg twice daily
2. Lifestyle modification program + linagliptin (2.5mg) and metformin (850mg) twice daily

on the following parameters, after 24 months of treatment:

1. Glucose metabolism, evaluated by the oral glucose tolerance
2. Insulin resistance, evaluated by the oral glucose tolerance in 100% of the patients and by hyperglycemic clamp in 10 % of the patients
3. Insulin secretion, evaluated by the oral glucose tolerance in 100% of the patients and by hyperglycemic clamp in 10 % of the patients
4. Pancreatic beta cell function, evaluated by the oral glucose tolerance in 100% of the patients and by hyperglycemic clamp in 10 % of the patients
5. Systemic inflammation and cardiovascular risk factors, evaluated by cytokines interlelukin-6 (IL6), C-reactive protein (PCR), and measurement of the intima media thickness by ultrasound.

All the patients will have a basal evaluation with an oral glucose tolerance test, lipid profile, body composition, and IMT measurement by ultrasonography; and 10 % will be invited for the hyperglycemic clamp. After the basal evaluation, if the patients result with IMPAIRED GLUCOSE TOLERANCE and have at least 2 risk factors, they will be invited to the intervention phase where they will be randomized to one of the two treatment groups.

Patients will have a follow-up visit every month to review the adherence to the lifestyle modification program and to the medication. Every 6 months OGTT will be performed on all the patients, and in a subset of patients hyperglycemic clamp will be performed at 0, 6 and 12 months. After 18 and 24 months, patients will repeat the same evaluation performed as the basal evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prediabetes, defined for the existence impaired glucose tolerance (Glucose between 140 and 199 mg/dL at the 2 hours of the Oral Glucose Tolerance test (OGTT) ) with or without impaired fasting glucose (Fasting glucose between 100 and 125 mg/dL)
* Patients who accept to participate in the study and sign the informed consent letter.

Exclusion Criteria:

* Patients with diagnosed Type 2 Diabetes Mellitus previously or detected during the OGTT
* Patients in actual treatment or during the last 3 months with metformin, pioglitazone or another antidiabetic drug, including insulin.
* Serum creatinine > 1.6 mg/dL
* Hypertriglyceridemia very high (>500 mg/dL)
* Pregnant women
* Altered arterial hypertension (Systolic > 180 mmHg or Diastolic >105 mmHg)
* Excessive alcohol intake, acute or chronic
* Medications or medical conditions that affect glucose homeostasis (thiazides, beta blockers, glucocorticoids for systemic use, weight-reducing drugs or anorexigenics, Cushing's syndrome, Thyrotoxicosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-01; Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change from basal fasting and post2h OGTT glucose levels at 12 and 24 months | 12 and 24 months
  Fasting and post-2h OGTT glucose values (mg/dl)

SECONDARY OUTCOMES:
Change from basal pancreatic beta cell function at 12 and 24 months | 12 and 24 months
  Evaluated with the measurements of glucose and insulin during the oral glucose tolerance test; as well as with the glucose and insulin measurements from the hyperglycemic clamp, as the Disposition index.
Change from basal insulin sensitivity at 12 and 24 months | 12 and 24 months
  Insulin sensitivity evaluated during the oral glucose tolerance test by the Matsuda index, and reported as an arbitrary units.
Change from basal Weight at 12 and 24 months | 12 and 24 months
  Weight measurement during the study, in kg
Incidence of type 2 diabetes | 24 months
  New reported cases with T2D according the the ADA diagnostic criteria

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Guardado-Mendoza, MDPhD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Faerch K, Borch-Johnsen K, Holst JJ, Vaag A. Pathophysiology and aetiology of impaired fasting glycaemia and impaired glucose tolerance: does it matter for prevention and treatment of type 2 diabetes? Diabetologia. 2009 Sep;52(9):1714-23. doi: 10.1007/s00125-009-1443-3. Epub 2009 Jul 10. PMID 19590846
- [Background] Faerch K, Vaag A, Holst JJ, Glumer C, Pedersen O, Borch-Johnsen K. Impaired fasting glycaemia vs impaired glucose tolerance: similar impairment of pancreatic alpha and beta cell function but differential roles of incretin hormones and insulin action. Diabetologia. 2008 May;51(5):853-61. doi: 10.1007/s00125-008-0951-x. Epub 2008 Mar 4. PMID 18317726
- [Background] Faerch K, Vaag A, Holst JJ, Hansen T, Jorgensen T, Borch-Johnsen K. Natural history of insulin sensitivity and insulin secretion in the progression from normal glucose tolerance to impaired fasting glycemia and impaired glucose tolerance: the Inter99 study. Diabetes Care. 2009 Mar;32(3):439-44. doi: 10.2337/dc08-1195. Epub 2008 Dec 3. PMID 19056613
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Chiasson JL, Josse RG, Gomis R, Hanefeld M, Karasik A, Laakso M; STOP-NIDDM Trail Research Group. Acarbose for prevention of type 2 diabetes mellitus: the STOP-NIDDM randomised trial. Lancet. 2002 Jun 15;359(9323):2072-7. doi: 10.1016/S0140-6736(02)08905-5. PMID 12086760
- [Background] Drucker DJ, Sherman SI, Gorelick FS, Bergenstal RM, Sherwin RS, Buse JB. Incretin-based therapies for the treatment of type 2 diabetes: evaluation of the risks and benefits. Diabetes Care. 2010 Feb;33(2):428-33. doi: 10.2337/dc09-1499. No abstract available. PMID 20103558
- [Background] Rosenstock J, Klaff LJ, Schwartz S, Northrup J, Holcombe JH, Wilhelm K, Trautmann M. Effects of exenatide and lifestyle modification on body weight and glucose tolerance in obese subjects with and without pre-diabetes. Diabetes Care. 2010 Jun;33(6):1173-5. doi: 10.2337/dc09-1203. Epub 2010 Mar 23. PMID 20332357
- [Background] Kim SH, Liu A, Ariel D, Abbasi F, Lamendola C, Grove K, Tomasso V, Reaven G. Pancreatic beta cell function following liraglutide-augmented weight loss in individuals with prediabetes: analysis of a randomised, placebo-controlled study. Diabetologia. 2014 Mar;57(3):455-62. doi: 10.1007/s00125-013-3134-3. Epub 2013 Dec 11. PMID 24326527
- [Background] Heise T, Graefe-Mody EU, Huttner S, Ring A, Trommeshauser D, Dugi KA. Pharmacokinetics, pharmacodynamics and tolerability of multiple oral doses of linagliptin, a dipeptidyl peptidase-4 inhibitor in male type 2 diabetes patients. Diabetes Obes Metab. 2009 Aug;11(8):786-94. doi: 10.1111/j.1463-1326.2009.01046.x. Epub 2009 May 19. PMID 19476474
- [Background] Craddy P, Palin HJ, Johnson KI. Comparative effectiveness of dipeptidylpeptidase-4 inhibitors in type 2 diabetes: a systematic review and mixed treatment comparison. Diabetes Ther. 2014 Jun;5(1):1-41. doi: 10.1007/s13300-014-0061-3. Epub 2014 Mar 25. PMID 24664619
- [Background] Del Prato S, Taskinen MR, Owens DR, von Eynatten M, Emser A, Gong Y, Chiavetta S, Patel S, Woerle HJ. Efficacy and safety of linagliptin in subjects with type 2 diabetes mellitus and poor glycemic control: pooled analysis of data from three placebo-controlled phase III trials. J Diabetes Complications. 2013 May-Jun;27(3):274-9. doi: 10.1016/j.jdiacomp.2012.11.008. Epub 2013 Feb 9. PMID 23403068

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03004612/Prot_SAP_000.pdf